CLINICAL TRIAL: NCT06380309
Title: An Open Label, Dose-escalation and Extension, Phase I Clinical Study on Evaluating Safety, Tolerability and Pharmacodynamics of Intravenous Administration of IDOV-SAFE in Patients With Advanced Malignant Solid Tumors Who Have Failed in Standard Treatment.
Brief Title: A Clinical Study on Evaluating Intravenous Administration of IDOV-SAFE
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Chief of Beijing Cancer Hospital, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY001-I001
Record Dates: First submitted 2024-04-15; First posted 2024-04-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Advanced Malignant Solid Tumor of Digestive System

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- IIA1：1E9 PFU of oncolytic virus, sequentially combination (Experimental): Subjects with MSS colorectal cancer was recruited to this Arm.Intravenous injection of 1E9 PFU oncolytic virus, following disease progression on IDOV-SAFETM monotherapy, combination therapy with IDOV-SAFETM, toripalimab, and fruquintinib was administered.
  Interventions: Biological: IIA1：1E9 PFU of oncolytic virus, sequentially combination
- IIA2：3E9 PFU of oncolytic virus, sequentially combination (Experimental): Subjects with MSS colorectal cancer was recruited to this Arm.Intravenous injection of 3E9 PFU oncolytic virus, following disease progression on IDOV-SAFETM monotherapy, combination therapy with IDOV-SAFETM, toripalimab, and fruquintinib was administered.
  Interventions: Biological: IIA2：3E9 PFU of oncolytic virus, sequentially combination
- IIC1：1E9 PFU of oncolytic virus, early combination (Experimental): Subjects with MSS colorectal cancer was recruited to this Arm.Intravenous injection of 1E9 PFU oncolytic virus, following treatment with IDOV-SAFETM, subjects received combination therapy with IDOV-SAFETM, toripalimab, and fruquintinib starting from cycle 2 or cycle 3.
  Interventions: Biological: IIC1：1E9 PFU of oncolytic virus, early combination
- IIC2：3E9 PFU of oncolytic virus, early combination (Experimental): Subjects with MSS colorectal cancer was recruited to this Arm.Intravenous injection of 3E9 PFU oncolytic virus, following treatment with IDOV-SAFETM, subjects received combination therapy with IDOV-SAFETM, toripalimab, and fruquintinib starting from cycle 2 or cycle 3.
  Interventions: Biological: IIC2：3E9 PFU of oncolytic virus, early combination
- IID：3E9 PFU of oncolytic virus, Immuno-Oncology free combination (Experimental): Subjects with MSS colorectal cancer was recruited to this Arm. After one cycle of IDOV-SAFETM treatment of 3E9 PFU, subjects received combination therapy with IDOV-SAFETM and fruquintinib starting from cycle 2.
  Interventions: Biological: IID：3E9 PFU of oncolytic virus, Immuno-Oncology free combination
- IIB：Other Gastrointestinal tumors (Experimental): Patients with digestive system tumors, such as cholangiocarcinoma, gastric cancer, esophageal squamous cell carcinoma, and hepatocellular carcinoma, received combination therapy with IDOV-SAFE + Toripalimab + Fruquintinib after progression on IDOV-SAFETM monotherapy.
  Interventions: Biological: IIB：Other Gastrointestinal tumors

INTERVENTIONS:
Biological: IIA1：1E9 PFU of oncolytic virus, sequentially combination — Intravenous injection of 1E9 PFU oncolytic virus, following disease progression on IDOV-SAFETM monotherapy, combination therapy with IDOV-SAFETM, toripalimab, and fruquintinib was administered.
  Arms: IIA1：1E9 PFU of oncolytic virus, sequentially combination
Biological: IIA2：3E9 PFU of oncolytic virus, sequentially combination — Intravenous injection of 3E9 PFU oncolytic virus, following disease progression on IDOV-SAFETM monotherapy, combination therapy with IDOV-SAFETM, toripalimab, and fruquintinib was administered.
  Arms: IIA2：3E9 PFU of oncolytic virus, sequentially combination
Biological: IIC1：1E9 PFU of oncolytic virus, early combination — Intravenous injection of 1E9 PFU oncolytic virus, following treatment with IDOV-SAFETM, subjects received combination therapy with IDOV-SAFETM, toripalimab, and fruquintinib starting from cycle 2 or cycle 3.
  Arms: IIC1：1E9 PFU of oncolytic virus, early combination
Biological: IIC2：3E9 PFU of oncolytic virus, early combination — Intravenous injection of 3E9 PFU oncolytic virus, following treatment with IDOV-SAFETM, subjects received combination therapy with IDOV-SAFETM, toripalimab, and fruquintinib starting from cycle 2 or cycle 3.
  Arms: IIC2：3E9 PFU of oncolytic virus, early combination
Biological: IID：3E9 PFU of oncolytic virus, Immuno-Oncology free combination — After one cycle of IDOV-SAFETM treatment of 3E9 PFU, subjects received combination therapy with IDOV-SAFETM and fruquintinib starting from cycle 2.
  Arms: IID：3E9 PFU of oncolytic virus, Immuno-Oncology free combination
Biological: IIB：Other Gastrointestinal tumors — combination therapy with IDOV-SAFE + Toripalimab + Fruquintinib after progression on IDOV-SAFETM monotherapy.
  Arms: IIB：Other Gastrointestinal tumors

SUMMARY:
Subjects were Chinese patients with histologically or cytologically confirmed advanced malignant solid tumors (mainly focused on MSS type colon and rectal cancer) who had failed standard systemic therapy and were inoperable.

The first stage was the dose escalation stage, which was divided into 4 dose groups according to the "3+3" dose escalation principle. One patient was enrolled in the first dose group, and 3-6 patients were enrolled in each of the latter three dose groups, with a total of 10-19 patients enrolled.

The second stage is the security extension stage, which is selected by SMC 1-2 dose cohorts were expanded for safety and divided into three cohorts in total(IIA, IIB, IIC) to explore the safety of sequential or combined administration modes with immune targeted therapy. Each cohort included 6-12 subjects at different dose levels, and three cohorts could be carried out at the same time.

The third stage is the dose expansion stage. According to the safety, PK and clinical data of the three cohorts in the second stage, 1-2 cohorts were selected by SMC for dose expansion. The sample size of each cohort was expanded to 20 cases on the original basis. The estimated ORR of the trial drug was 24%, and the ORR of the standard treatment was 5%. When the type I error was one-sided 0.025, and the power was 80%, the sample size was estimated by the normal approximation method. So each dose expansion phase A minimum of 20 subjects were required to be enrolled in the cohort.

DETAILED DESCRIPTION:
Overview of clinical trial The therapeutic dose in mice was 1x108 PFU, and the maximum starting dose in humans was 2.67x10^9 PFU according to the "Guidelines for the estimation of the maximum recommended starting dose of drugs in the First clinical trial of Healthy Adult Volunteers".

Phase 1: Dose escalation phase:

We plan to enroll 10 to 19 patients in China with histologically or cytologically confirmed advanced solid tumors who have failed to respond to standard treatment or have no standard treatment options for IDOV-SAFETM intravenous administration. Patients with MSS colorectal cancer were included in this stage.

This phase included four dose groups of 1x10^9 PFU, 3x10^9 PFU, 1x10^10 PFU and 3x10^10 PFU. One subject was enrolled in the first dose group, and the other dose groups were increased by a "3+3" method, with 3-6 subjects in each group. All participants in each dose arm could not be escalated to the next dose arm until they had completed the 21-day safety assessment.

Dose escalation or Settings may be adjusted at the discretion of the Safety Committee (SMC).

Phase 2: Security Extension Phase:

One or two dose levels determined by MTD or SMC were selected for expansion. This phase was divided into four cohorts,:

Cohort IIA: Patients with MSS colorectal cancer who progressed after IDOV-SAFETM monotherapy were treated with IDOV-SAFETM+ toripalimab-furoquininib combination therapy

IIA1: Approximately 6~12 subjects were enrolled in the first dose group. IIA2: About 6~12 subjects were enrolled in the second dose group;

Cohort IIB: Patients with cholangiocarcinoma, gastric cancer, esophageal squamous cell carcinoma, liver cancer and other digestive system tumors were enrolled.

Enroll 6-12 subjects in the second dose group;

Cohort IIC: patients with MSS colorectal cancer were enrolled. After 2 cycles of IDOV-SAFETM treatment, the subjects were treated with IDOV-SAFETM, toripalimab and fuquinitinib combination therapy.

IIC1: Approximately 6~12 subjects were enrolled in the first dose group. IIC2: About 6~12 subjects were enrolled in the second dose group;

ⅡD：Patients with MSS-type colorectal cancer were included. After one cycle of IDOV-SAFETM treatment, combined therapy with IDOV-SAFETM and fruquintinib was initiated starting from the second cycle.

About 6~12 subjects were enrolled in the second dose group;

Phase III: Dose expansion phase:

According to the safety, PK and clinical data of the four cohorts in the second phase, one or two cohorts were selected by SMC for dose expansion, and the sample size of each cohort was expanded to 20 cases.

After completing the first cycle of dosing, all subjects received subsequent cycles of dosing after 21 days of safety assessment. The course of treatment, related examinations and tumor efficacy evaluation were consistent between the monotherapy phase and the combination phase. The patients were treated with intravenous injection on D1, 3 and 5 of each course of treatment according to every 3 weeks (21 days) as a course of treatment. Safety checks were performed for each cycle. Tumor efficacy was evaluated every 2 cycles (every 6 weeks) according to RECIST1.1 and iRECIST standards. Pharmacodynamic tests (including tumor markers, T cell subsets, cytokines, viral load in tumor tissue, etc.), viral distribution detection, and TCR-Seq detection were performed regularly.

When the subject met the 9.1 criteria for the end of treatment for the subject, the treatment period ended and the subject entered the long-term safety and survival follow-up period.

Long-term SAFETY AND SURVIVAL FOLLOW-UP:

Adverse events that occurred in each subject from the first dose of the study were collected throughout the course of the study, and long-term safety and survival follow-up was to continue for 2 years after the last dose (visits were performed every 8 weeks until death or loss to follow-up or the end of survival follow-up). Before the subjects started a new antineoplastic therapy, they were examined accordingly according to the "6.9 Clinical Trial Schedule". Survival was confirmed by telephone visits after the initiation of a new antineoplastic therapy.

Other medications:

If, according to the investigator's judgment during the trial, the patient is considered to be safe but not effective at the current dose, the subject needs to withdraw from the trial, and the trial SMC meeting has decided and the next (higher) dose group has been initiated. At the discretion of the investigator, the higher dose of the trial drug could be administered to the subject who was withdrawing from the trial.

In order to ensure the interests of the subjects to the greatest extent, after the end of the treatment, if the subjects are evaluated by the investigators and the subjects agree, this clinical trial can provide "compensatory medication", and provide IDOV-SAFETM to the subjects for free. At the same time, the patients need to sign the informed consent for the use of "compensatory medication".

ELIGIBILITY:
Inclusion Criteria:

1. Be fully aware of this study and voluntarily sign ICF. 2. Age range from 18 to 75 years old at the time of screening, gender is not limited.

3. At the time of screening, patients with advanced malignant digestive system tumors confirmed by histology or cytology, including MSS type colorectal cancer, bile duct cancer, stomach cancer, esophageal cancer, liver cancer, etc.

4. At the time of screening, the disease has progressed after or during standard treatment; Subjects with advanced malignant digestive system tumors with no standard treatment currently available, intolerance to chemotherapy, or greater than or equal to progression after 2-line system therapy.

1. Be fully aware of this study and voluntarily sign ICF.
2. Age range from 18 to 70 years old at the time of screening, gender is not limited.
3. At the time of screening, patients with advanced malignant digestive system tumors confirmed by histology or cytology, including MSS type colorectal cancer, bile duct cancer, stomach cancer, esophageal cancer, liver cancer, etc.
4. At the time of screening, the disease has progressed after or during standard treatment; Subjects with advanced malignant digestive system tumors with no standard treatment currently available, intolerance to chemotherapy, or greater than or equal to progression after 2-line system therapy.
5. When screening, the ECOG score of physical strength score is 0 or 1.
6. Life expectancy assessed by the investigator at the time of screening was ≥3 months.
7. Subjects had adequate organ function at baseline:

   a) Bone marrow function (no growth factor support therapy or component transfusion within 14 days prior to screening) : i. Neutrophil absolute value (ANC) ≥1.5×109/L; ii. Hemoglobin (HB) ≥90g/L; iii. Platelet count (PLT) ≥75×109/L; b) Liver function: i. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 times the upper limit of normal (ULN) (ALT and AST≤ 3 times ULN for liver metastasis or hepatocellular carcinoma); ii. Total blood bilirubin ≤ 1.5 ULN (in subjects with liver metastasis or hepatocellular carcinoma or Gilbert syndrome or familial benign nonbinding hyperbilirubinemia, the acceptable range of this indicator is ≤2.5 ULN); c) Renal function: serum creatinine ≤ 1.5x ULN or creatinine clearance ≥50mL/min;
8. Fertile female subjects must have negative blood beta-HCG test results within 7 days prior to enrollment.
9. Subjects must agree to use highly effective contraception for at least 90 days from the start of the ICF to the end of the study.
10. At least one measurable lesion according to RECIST v1.1 criteria, The target lesion had not been treated with radiotherapy or had definite radiographic progression after previous radiotherapy.

Exclusion Criteria:

1. At the time of screening, advanced malignant tumors have a chance of being cured by radical treatment.
2. Asymptomatic brain metastases such as untreated ones at the time of screening; Subjects with symptomatic central nervous system (CNS) metastatic or cancerous meningitis; Or there was other evidence of uncontrolled central nervous system or meningeal metastases in subjects who were judged by the investigator to be unsuitable for enrollment.
3. Prior to enrollment, there was severe chronic or active infection: active hepatitis B (HbsAg positive, HBV DNA test value greater than the upper limit of normal); Active hepatitis C (those with positive anti-HCV antibodies are further tested positive for HCV RNA); A known history of immunodeficiency virus (HIV) disease or a positive HIV antibody test; Other conditions requiring systemic anti-infective treatment in the 4 weeks prior to initial use of the investigational drug include, but are not limited to, hospitalization for infectious complications, bacteremia, severe pneumonia, or active tuberculosis.
4. At the time of screening, patients had a history of active autoimmune diseases such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc., or were receiving long-term systemic steroids (prednisone >10mg/ day or equivalent doses of the same drug) or any other form of immunosuppressant therapy within 14 days prior to the first use of the study drug.
5. Have received allogeneic tissue or solid organ transplantation.
6. There is evidence of clinically significant immunodeficiency, such as primary immunodeficiency status, such as severe combined immunodeficiency disease (SCID); Combined with opportunistic infections.
7. Anticoagulants or antiplatelet drugs should be used before injection and should not be interrupted, including: aspirin should not be stopped within 7 days before injection; Coumarin that cannot be stopped within 7 days prior to injection; Direct thrombin inhibitors (such as dabigatrun) or direct factor Xa inhibitors (such as rivaroxaban, apixaban, and neperoxaban) that cannot be discontinued within 4 days prior to injection; Low molecular weight heparin (LMWH) should not be stopped within 24 hours before injection, and ordinary heparin (UFH) should not be stopped more than 4 hours before injection.
8. Have a history of severe cardiovascular and cerebrovascular disease, including but not limited to: congestive heart failure ≥II heart function grade of the New York Heart Association (NYHA); Left ventricular ejection fraction (LVEF) <50%; QT interval (QTcF) >470ms as corrected by the Fridericia method or prolonged QT interval syndrome; Acute coronary syndrome, aortic dissection, severe arrhythmia, stroke, or other grade 3 or higher cardiovascular and cerebrovascular events occurred within 6 months before first administration; The presence of uncontrolled hypertension (systolic blood pressure >140mmHg or diastolic blood pressure >90mmHg). Subjects with a history of hypertension are admitted to the study if their blood pressure is controlled below this standard and maintained with antihypertensive therapy.
9. Received treatment with other methods, including but not limited to chemotherapy, radiotherapy, biotherapy, endocrine therapy, immunotherapy, etc., within 4 weeks prior to the first use of the investigational drug.
10. Other diseases or abnormalities assessed by the investigator as unsuitable for participation in the study.
11. Vaccination against smallpox or monkeypox within 10 years before the first use of study drug.
12. Allergy to macromolecular antibody drugs or small molecule TKI drugs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2024-05-06 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence of dose-limiting toxicity (DLT) | 21 days after the administration, up to 2 months
  Occurrence of dose-limiting toxicity (DLT) on dose escalation phase
Incidence of adverse events (AE) | After the subject completed the study, about 1 year
  Incidence of adverse events (AE) in monotherapy and combination phase
The objective response rate (ORR) from baseline (data on screenning) for IDOV-Safe under three different combination regimens. | After subject complete tumor assessment, about half a year
  The objective response rate (ORR) from baseline (data on screenment) for IDOV-Safe under three different combination regimens.

SECONDARY OUTCOMES:
The level of (non-essential) viral DNA in tumor tissue | After the subject completed the treatment, about 1 year
  The investigator will select the subjects suitable for tumor tissue sample collection, with their informed consent.
Tumor markers | Every 6 weeks during screening and continued treatment, about 1 year
  Tumor marker test was performed every 6 weeks during screening and continued treatment
Anti-vaccinia virus neutralizing antibody test(VV-Nab) | After the subject completed the treatment, about 1 year
  Peripheral blood samples were collected for vaccinia virus neutralizing antibody (VV-Nab) detection at 0h (-60min) before the first dose on D1 and on D7 ± 1d after the first dose on D1. For subsequent cycles, samples were only collected at 0h (-60min) before the dose on D1.
Levels of viral DNA in blood | After the subject completed the treatment, about 1 year
  During the dose escalation phase, expansion phase and dose expansion phase, peripheral blood samples were collected at 25 time points: 2 hours before each injection of D1, D3 and D5, and 30 minutes ± 5 minutes, 2 hours ± 15 minutes, 4 hours ± 30 minutes, 8 hours ± 1 hour, 12 hours ± 1 hour, 24 hours ± 1 hour, 36 hours ± 2 hours after each injection, as well as 48 hours ± 2 hours after the last injection of D5. In the second and third cycles, peripheral blood samples were collected at 6 time points: 2 hours before each injection of D1 and 30 minutes ± 5 minutes, 2 hours ± 15 minutes, 8 hours ± 1 hour, 12 hours ± 1 hour, 24 hours ± 1 hour after each injection. In the second and third cycles, peripheral blood samples were collected at 2 time points: 2 hours before each injection of D3 and D5 and 30 minutes ± 5 minutes after each injection. Viral DNA and live virus load were measured in all samples, and the half-life was calculated.
Levels of viral DNA in saliva | Before and 2±1 h after administration, up to 31 days
  Saliva was collected before and 2±1 h after administration for comparison
T cell subsets | Screening period and 24 hours ±4 hours after the first administration, D4±1d, D7±1d, and every 6 weeks during the continuous treatment period, about 1 year
  T cell subsets were evaluated four times during the screening period and 24 hours ±4 hours after the first administration, D4±1d, D7±1d, and every 6 weeks during the continuous treatment period
Cytokines | Screening stage and D7±1d after the first dose, and every 6 weeks during the continuous treatment period, about 1 year
  Cytokines were evaluated at the screening stage and D7±1d after the first dose, and every 6 weeks during the continuous treatment period
Combine ORR | Every 6 weeks (±7 days) after initial administration, about 1 year
  Under the sequential treatment regimen, the combined ORR of the combination therapy was evaluated using the time of disease progression on monotherapy as the baseline.
DCR | Every 6 weeks (±7 days) after initial administration, about 1 year
  The sum of the proportion of subjects with CR 、PR or SD
DOR | Every 6 weeks (±7 days) after initial administration, about 1 year
  The time between the start of the first assessment of the tumor as CR or PR and the second assessment as PD(Progressive Disease) or death from any cause
PFS | Every 6 weeks (±7 days) after initial administration, about 1 year
  The time, measured in days, from the date of first treatment to disease progression or death from any cause. Disease progression and death were measured in terms of preoccurrence. Progression included radiographic progression or clinical progression as assessed by the investigator.
OS | Every 6 weeks (±7 days) after initial administration, about 5 years
  The time from the date of first treatment to death from any cause, measured in days
PFS2 | Every 6 weeks (±7 days) after initial administration, about 1 year
  Progression-free survival until second disease progression or death

OTHER OUTCOMES:
Exploratory endpoint | After the subject completed the study, about 1 year
  Dynamic changes in biomarkers (e.g., CD4, CD8, PD-L1) in tissue specimens monitored before and after treatment.
Exploratory endpoint | After the subject completed the study, about 1 year
  Single-cell/spatial transcriptomic/TCR sequencing was utilized to investigate changes in the tumor microenvironment and peripheral blood immune profiles.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, PHD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No